CLINICAL TRIAL: NCT00096967
Title: An Open-Label, Multicenter Extension Study of rhuMAb VEGF (Bevacizumab) in Subjects Treated in a Previous Genentech-Sponsored Cancer Study
Brief Title: A Study to Evaluate Avastin in Patients Treated in a Previous Genentech-Sponsored Cancer Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: AVF2540g; NCT00066560 (obsolete NCT alias)
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer; Colorectal Cancer; Metastases
Keywords: Metastatic breast cancer; Metastatic colorectal cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab

INTERVENTIONS:
Drug: Avastin (bevacizumab)

SUMMARY:
This is a multicenter, open-label extension study. Subjects who have received rhuMAb VEGF therapy in Study AVF2107g, AVF2119g, or AVF2192g and who completed the parent study are eligible for inclusion in this trial. Subjects who have received placebo in Study AVF2107g or AVF2192g are also eligible.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Previous participation in and completion of one of the following Genentech-sponsored rhuMAb VEGF Phase II or Phase III cancer studies: AVF2107g, AVF2119g, or AVF2192g
* Use of an effective means of contraception in men and in women of childbearing potential
* For subjects who received placebo in the parent study, current antitumor therapy not exceeding third-line treatment for disease progression

Exclusion Criteria:

* Compromised renal or hepatic function, as defined in the parent protocol
* EGOG status of 3 or greater
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored rhuMAb VEGF cancer study
* ANC of <1500/uL
* Platelet count of <75,000/uL
* International normalized ration (INR) >=1.5 (except those subjects who have been given approval to receive full-dose warfarin plus rhuMAb VEGF)
* Total bilirubin of >1.6 mg/dL for patients receiving irinotecan, for all others total bilirubin of >2.0 mg/dL
* AST or ALT >5 times upper limit of normal for subjects with documented liver metastases; >2.5 times the upper limit of normal for subjects without evidence of liver metastases
* Serum creatinine of >2.0 mg/dL
* Hemoglobin of <9 gm/dL (may be transfused or receive epoetin alfa [e.g., Epogen] to maintain or exceed this level)
* Inability to comply with study and/or follow-up procedures
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
* Any unresolved or irreversible rhuMAb VEGF-related ongoing serious adverse event occurring during the parent study
* Clinically significant cardiovascular disease (e.g., uncontrolled hypertension [blood pressure of >160/110 mmHg on medication], previous myocardial infarction, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac dysrhythmia requiring medication, or peripheral vascular disease (Grade II or greater)
* History or evidence upon physical examination of CNS disease (e.g., primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of stroke)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study
* Fine needle aspirations or core biopsies within 7 days prior to Day 0
* Chronic, daily treatment with aspirin (>325 mg/day) or nonsteroidal anti inflammatory medications (of the kind known to inhibit platelet function at doses used to treat chronic inflammatory diseases)
* Pregnancy (positive pregnancy test) or lactation
* Proteinuria at baseline or clinically significant impairment of renal function
* Serious, nonhealing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2002-10; Study Completion 2004-07 (Actual)